CLINICAL TRIAL: NCT02765464
Title: Predicting Acute Kidney Injury in Critically Ill Trauma Patients Using Metalloproteinase 2 (TIMP2) and Insulin-like Growth Factor Binding Protein7 (IGFBP 7)
Brief Title: Acute Kidney Injury in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Ronak Raval, MD, Loma Linda University
Other Study IDs: 5160026
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Acute Renal Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute kidney injury (AKI) in critically ill trauma patients has been shown to significantly increase mortality, length of stay, and costs, however detection has proven difficult as markers like elevated creatinine and decreased urine output may take days to manifest and are late indicators of AKI. The combination of two urinary biomarkers, Tissue Inhibitor of Metalloproteinase 2 (TIMP-2) and Insulin-like Growth Factor Binding Protein 7 (IGFBP-7), has been shown to increase within 12 hours following renal insult, allowing assessment of risk for developing acute kidney injury. Therefore, the investigators plan to assess if acute kidney injury in critically ill trauma patients can be determined earlier using urinary TIMP-2 and IGFBP-7 via the NephroCheck testing system. These markers have not been specifically evaluated in trauma patients at risk of AKI.

ELIGIBILITY:
Inclusion Criteria:

* trauma patients with multiple injuries;
* abdominal injuries;
* crush injuries;
* those who present in shock (systolic blood pressure <90 or mean arterial pressure <65);
* require blood transfusions, vasopressors or mechanical ventilation

Exclusion Criteria:

* known pregnancy;
* patients under 21 years of age;
* known moderate to severe AKI prior to enrollment and end stage renal disease. known moderate to severe AKI prior to enrollment and end stage renal disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be trauma patients with multiple injuries.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Measurement of u rinary metalloproteinase 2 (TIMP-2) and Insulin-like growth factor binding protein 7 (IGFBP-7) biomarker elevation that corresponds to acute kidney injury by creatinine and urine output | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Raval, MD, Principal Investigator — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No